CLINICAL TRIAL: NCT03103425
Title: Evaluation of StatNet Device for EEG Recordings
Brief Title: Evaluation of StatNet Device for Electroencephalogram (EEG) Recordings
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: HydroDot, Inc. (Industry)
Responsible Party: Principal Investigator, Trudy Pang, Instructor in Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2009P000058
Record Dates: First submitted 2009-06-26; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy; Seizures
Keywords: New onset seizures
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to develop an emergency electroencephalogram (EEG) device, StatNet, that can be placed quickly by minimally-trained personnel and interpreted remotely for rapid identification of seizures.

ELIGIBILITY:
Inclusion Criteria:

* Adults > age 18
* Epileptiform discharges present on routine EEG

Exclusion Criteria:

* Open head wounds
* Medically Unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients Inpatients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States